CLINICAL TRIAL: NCT01288859
Title: Physiological Effects of New Polyphenol-enriched Foods in Healthy Humans
Brief Title: Physiological Effects of New Polyphenol-enriched Foods in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Vincenzo Fogliano, Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DSA-FF-01
Record Dates: First submitted 2011-01-27; First posted 2011-02-03 (Estimated); Results first posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: polyphenols; curcumin; bioavailability; cocoa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- encapsulated curcumin (Experimental)
  Interventions: Other: encapsulated curcumin
- encapsulated curcumin + PQG (Experimental): PQG means Piperine, Quercetin and Genistein
  Interventions: Other: encapsulated curcumin + PQG
- free cocoa polyphenol (Active Comparator)
  Interventions: Other: free cocoa polyphenol
- control (Placebo Comparator)
  Interventions: Other: control nut cream
- encapsulated cocoa polyphenols (Experimental)
  Interventions: Other: encapsulated cocoa polyphenols
- free curcumin (Active Comparator): Subjects will consume bread added with free curcumin
  Interventions: Other: free curcumin

INTERVENTIONS:
Other: free curcumin — free curcumin in bread, dosage 1g/100g, 200g/day per 1 day
  Arms: free curcumin
Other: encapsulated curcumin — encapsulated curcumin-enriched bread, 1g/100g bread, 200g bread/day
  Arms: encapsulated curcumin
Other: encapsulated curcumin + PQG — bread enriched with encapsulated curcumin plus piperine, quercetin and genistein, 1g/100g bread, 200g bread/day
  Arms: encapsulated curcumin + PQG
Other: free cocoa polyphenol — nut cream enriched with free cocoa polyphenols, 1,5 g/100g cream, 100g/day per 1 day
  Arms: free cocoa polyphenol
Other: encapsulated cocoa polyphenols — nut cream enriched with encapsulated cocoa polyphenols, 1,5 g/100g cream, 100g/day per 1 day
  Arms: encapsulated cocoa polyphenols
Other: control nut cream — nut cream, cocoa polyphenols 0g/100g cream, 100 g/day per 1 day
  Arms: control

SUMMARY:
Polyphenolic compounds exert several health benefits depending on bioavailability. Encapsulation may improve bioavailability of these compounds.This study will evaluate bioavailability of some polyphenols (curcumin and cocoa polyphenols) from new enriched-foods. In particular bread and nut based creams will be used as food matrices to include free or encapsulated polyphenols.

DETAILED DESCRIPTION:
Polyphenolic compounds are abundant in foods and have been suggested to exert several health benefits including prevention of cancer, cardiovascular disease, suppressing inflammation, diabetes, etc. These properties are mediated by bioavailability of individual polyphenols that is, in turn, influenced by food properties (food matrix, technological processing, etc.), interaction with other compounds, and host related factors. Some well-studied dietary polyphenols include catechins from tea, curcumin from turmeric, procyanidins and anthocyanidins in grapes, berries, and dark chocolate. These compounds have strong antioxidative activities in vitro and have been suggested to have several beneficial health effects.

Curcumin, a phenolic compound deriving from turmeric spice, shows many biological and pharmacological effects, and clinical studies in humans proved that it's extremely safe and well tolerated even at very high doses (8-12 g/day). However, curcumin has not yet been approved as a therapeutic agent, because of its very low bioavailability depending on a poor absorption, rapid metabolism and rapid systemic clearance. Different approaches have been investigated to improve curcumin bioavailability. Among them, the use of adjuvants that interferes with metabolic pathways of curcumin, like piperine, represents one of the main strategies used to enhance its bioavailability. A further approach consists on manufacturing of curcumin containing liposomes, phospholipids complexes or nanoparticles. For polymer-based nanoparticles, maintenance of biological activity, increased absorption and delayed delivery was reported.

Cocoa based products are widely consumed in many countries, and indications of health benefits by some cocoa constituents, mainly polyphenols, have also been reported. Cocoa contains very high levels of polyphenols, in particular flavanols and among these, mainly epicatechins. The bioavailability of cocoa polyphenols has been measured in several human studies from acute consumption of cocoa rich beverages or chocolate. Monomeric flavonoids as well as dimeric and trimeric procyanidins were detected in human plasma over 2-3 hours from consumption. Plasma concentration of cocoa polyphenols were often in the nanomolar or low micromolar range. Donovan and coworkers demonstrated that commercial available chocolate samples contain a predominance of the less bioavailable (-)-catechin enantiomer as compared to the (+)-catechin which is present in most other plant derived foods. This may explain the relatively low bioavailability of catechins from chocolate and cocoa-containing products. The food matrix seems to be an important factor that may affect the bioavailability of cocoa polyphenols. For instance, proteins in the food matrix are supposed to form highly polymerized complexes with procyanidins, which can reduce bioaccessibility of these phenolic compounds. However, the potential negative effect of protein content in foods was not confirmed in a study that evaluated the cocoa polyphenols bioavailability after the intake of a milk-powder cocoa beverage. However, concurrent carbohydrates consumption seems to increase significantly the uptake of flavonols in humans. Little is known whether and to what extent oligomeric procyanidins from cocoa are absorbed. However, the biological activity of procyanidins with high polymerization degree may be partly attributed to their colonic breakdown products, including phenolic acids.

Actually there is also a growing interest in other biological properties of phenolic compounds in addition to their antioxidant effects; particularly, some evidences suggest that certain dietary phenols may modulate metabolic homeostasis. This is the case of chlorogenic acids, that are reported to play a potential role in modifying the pattern of intestinal glucose uptake and of other flavonoids (quercetin, catechins) that may modulate activation of GLP-1 receptor, involved in modulation of insulin and glucagon secretion, gastric emptying, and appetite.

In this randomized, crossover trial, serum, urine and fecal concentrations of curcumin and cocoa polyphenols, their parental compounds, metabolites and phenolic acids, following a two day multi-dose administration with six food sources, will be measured. All volunteers will undergo to six interventions - bread enriched with three different forms of curcumin (free, encapsulated, and encapsulated plus piperine) and nut based creams enriched with cocoa polyphenols (free or encapsulated one) or control cream (without enrichment). A one-week wash-out period will be included between two sequential treatments. Blood, urine and feces will be collected at time 0 (baseline), 24, and 48 hours; further blood samples at 0.5, 1, 2, 4, 6 hours after consumption of the first meal, and urine samples at 2 hours time intervals up to 10 hours, will be collected too. In particular, area under the curve (AUC) of serum and urine concentrations of parental compounds and metabolites in the time interval 0-24 hours will be calculated as primary outcomes. In addition the amount of total polyphenols in fecal samples will be measured.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years old, male and female
* Healthy by medical assessment
* Normal weight: BMI 18 - 25
* Sign of a written informed consent

Exclusion Criteria:

* Age > 18 and < 45 years old
* Pregnancy or breastfeeding
* Intestinal or metabolic diseases/disorders such as diabetic, renal, hepatic, hypertension, pancreatic or ulcer, including lactose-intolerance
* Previous abdominal/gastrointestinal surgery
* Regular consumption of medication
* Antibiotic therapy within 2 months previous the study
* Food allergies and intolerances (celiac disease, lactose intolerance, nut allergy etc)
* Unwilling to consume experimental foods
* Concurrent participation or having participated to another clinical trial during the last 3 weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Fogliano, Professor, Principal Investigator — University of Naples; Paola Vitaglione, Researcher, Study Director — University of Naples
Locations (1):
- Department of Food Science, Portici, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was performed at the ambulatory of Department of Food Science (University of Naples) among students of Agriculture Faculty. It began on December 2010 up to February 2011.
Pre-assignment Details: Subjects were enrolled after signing a Consent Form and were randomized to the treatments. All subjects enrolled completed the study.
Groups:
- Encapsulated Curcumin: Subjects consumed 2 bread portions/day of bread enriched with micro-encapsulated curcumin(1g/100g portion, i.e. 2g/day)
- Encapsulated Curcumin + PQG: Subjects consumed 2 bread portions/day of bread enriched with micro-capsules containing curcumin at dosage of 1 g/100 g plus 0.1% of Piperine, Quercetin and Genistein (PQG) (2g curcumin + 0.2g PQG/day) for one day.
- Free Cocoa Polyphenol: Subjects consumed 3 nut cream portions (33g each) enriched with cocoa polyphenols at dosage of 1.5g/day.
- Control Cream: Subjects consumed 3 nut cream portions (33g each).
- Encapsulated Cocoa Polyphenols: Subjects consumed 3 nut cream portions (33g each) enriched with encapsulated cocoa polyphenols at dosage of 1.5g/day.
- Free Curcumin: Subjects consumed 2 portions of bread enriched with free curcumin (1g/100g portion, i.e. 2g/day)
Period: Free Then Encapsulated Curcumin (1 Day)
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 5 | 0 | 0 | 0 | 0 | 5
Completed | 5 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 5 | 0 | 0 | 0 | 0 | 5
Completed | 5 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Encapsulated Then Free Curcumin (1 Day)
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 5 | 0 | 0 | 0 | 0 | 5
Completed | 5 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 5 | 0 | 0 | 0 | 0 | 5
Completed | 5 | 0 | 0 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Enc Curc + PQG Then Free Polyph. (1 Day)
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 0 | 5 | 5 | 0 | 0 | 0
Completed | 0 | 5 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 0 | 5 | 5 | 0 | 0 | 0
Completed | 0 | 5 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Free Polyph. Then Enc Curc + PQG (1 Day)
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 0 | 5 | 5 | 0 | 0 | 0
Completed | 0 | 5 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 0 | 0 | 0 | 5 | 5 | 0
Completed | 0 | 0 | 0 | 5 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Enc Polyph. Then Control Cream (1 Day)
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 0 | 0 | 0 | 5 | 5 | 0
Completed | 0 | 0 | 0 | 5 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 0 | 0 | 0 | 5 | 5 | 0
Completed | 0 | 0 | 0 | 5 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Control Cream Then Enc Polyph. (1 Day)
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Started | 0 | 0 | 0 | 5 | 5 | 0
Completed | 0 | 0 | 0 | 5 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants followed all the periods
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  Italy | 10

OUTCOME MEASURES:

1. Primary Outcome: Serum Polyphenol Concentrations Over 24h From Food Consumption
Description: Area Under the Curves (AUC) from 0 to 24h of parent polyphenols was calculated using a trapezoidal rule applied to the concentration-time curves of compounds.
Time Frame: 0, 0.5, 1, 2, 4, 6, and 24 hours post-dose
Population: The number of subjects was based on power calculations derived from our previous study. We calculated that, at α = 0.05 with a power of 80%, 8 subjects would allow us to detect a 20% difference in serum and urinary concentrations of parental compounds, glucuronides and phenolic acids.
Measure: Mean (Standard Error); unit: nmol*h/L
Groups:
- Free Curcumin: subjects consumed bread enriched with free curcumin
- Encapsulated Curcumin: subjects consumed bread enriched with encapsulated curcumin
- Encapsulated Curcumin + PQG: subjects consumed bread enriched with encapsulated curcumin plus piperine, quercetin and genistein
- Control Cream: subjects consumed cocoa-nut cream
- Free Cocoa Polyphenols: subjects consumed cocoa-nut cream enriched with cocoa polyphenols in the free form
- Encapsulated Cocoa Polyphenols: subjects consumed cocoa-nut cream enriched with encapsulated cocoa polyphenols
Arm/Group | Free Curcumin | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Control Cream | Free Cocoa Polyphenols | Encapsulated Cocoa Polyphenols
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
nmol*h/L | 1.7 (0.1) | 12.1 (1.1) | 7.7 (1.8) | 0.01 (0.00) | 7.3 (0.9) | 0.5 (0.1)
Statistical Analysis 1: Comparison: Free Curcumin vs Encapsulated Curcumin vs Encapsulated Curcumin + PQG vs Control Cream vs Free Cocoa Polyphenols vs Encapsulated Cocoa Polyphenols; Test type: Non-Inferiority or Equivalence — The results from LC-MS/MS analysis of parent polyphenols were analyzed and expressed as the absolute changes from the baseline to reduce possible effects of inter-subject fasting variability; p = 0.02, ANOVA; Mean Difference (Final Values) = 1, Standard Error of Mean 0.1

2. Primary Outcome: Urinary Excretion of Total Polyphenols
Description: Area Under the Curve (AUC) from 0 to 24h of total polyphenols (sum of parent polyphenols and metabolites)was calculated using a trapezoidal rule applied to the urinary concentration-time curves of compounds.
Time Frame: Time intervals: 0-2, 2-4, 4-6, 6-8, 10-24 hours post-dose.
Population: Basing on power analysis calculation on a previous work
Measure: Mean (Standard Error); unit: nmol•h/L
Groups:
- Encapsulated Curcumin: subjects consumed bread containing encapsulated curcumin
- Encapsulated Curcumin + PQG: subjects consumed bread containing encapsulated curcumin plus PQG (i.e. Piperine, Quercetin and Genistein)
- Free Cocoa Polyphenol: subjects consumed nut creams added with cocoa polyphenols
- Control: Subjects consumed white bread or nut cream
- Encapsulated Cocoa Polyphenols: subjects consumed nut creams added with encapsulate cocoa-polyphenols
- Free Curcumin: Subjects consumed bread added with free curcumin
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control | Encapsulated Cocoa Polyphenols | Free Curcumin
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
nmol•h/L | 2.0 (0.8) | 2.21 (1.27) | 9.67 (6.7) | 19.1 (12.3) | 4.92 (3.36) | 1.31 (0.81)
Statistical Analysis 1: Comparison: Encapsulated Curcumin vs Encapsulated Curcumin + PQG vs Free Cocoa Polyphenol vs Control vs Encapsulated Cocoa Polyphenols vs Free Curcumin; Statistical analysis was performed using the statistical package SPSS for Windows (version15). By the analysis of variance (ANOVA) for repeated measures the subjective time curves for all measured compounds were compared and tested for the effect of treatment and of time as factors. For all tests, following a significant main effect in the ANOVA, individual means were compared using the Bonferroni test (p < 0.05). Results were considered significant at p < 0.05; Test type: Superiority or Other; p = 0.01, ANOVA; Mean Difference (Final Values) = 0.9, Standard Error of Mean 0.01

3. Primary Outcome: Amount of Total Fecal Polyphenols
Description: Amount of parent polyphenols and metabolites in feces was calculated by multiplying net concentrations by the amount of feces.
Time Frame: 0 and 24 hours post-dose.
Measure: Mean (Standard Error); unit: nmol
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control | Encapsulated Cocoa Polyphenols | Free Curcumin
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
nmol | 3.49 (2.13) | 0.49 (0.01) | 27.98 (13.97) | 4.27 (4.52) | 150.97 (54.65) | 0.59 (0.38)
Statistical Analysis 1: Comparison: Encapsulated Curcumin vs Encapsulated Curcumin + PQG vs Free Cocoa Polyphenol vs Control vs Encapsulated Cocoa Polyphenols; Test type: Superiority or Other; p = 0.04, ANOVA; Mean Difference (Final Values) = 0.2, Standard Error of Mean 0.01

ADVERSE EVENTS:
Arm/Group | Encapsulated Curcumin | Encapsulated Curcumin + PQG | Free Cocoa Polyphenol | Control Cream | Encapsulated Cocoa Polyphenols | Free Curcumin
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes